CLINICAL TRIAL: NCT06078722
Title: Evaluation of the Effectiveness of the Use of a Carnitine-Orotate Complex and Biphenyl Dimethyl Dicarboxylate in the Pathogenetic Therapy of Metabolic-associated Fatty Liver Disease: a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kazakh Association of Internal Medicine Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: KAIMS-01
Record Dates: First submitted 2023-09-25; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Metabolic-associated Fatty Liver Disease (MAFLD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Cohort: Patients taking Carnitine-Orotate Complex and BDD regardless of study participation. The duration of observation for taking COCs and BDD is 6 months, and the duration of follow-up is 6 months.
- Control cohort: Patients who do not take Carnitine-Orotate Complex and BDD, regardless of study participation. Duration of patient observation - 12 months.

SUMMARY:
The goal of this observational study is to learn the effectiveness and safety of the use of Carnitine-Orotate Complex and Biphenyl Dimethyl Dicarboxylate in the pathogenetic therapy of metabolic-associated fatty liver disease (MAFLD)

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 18 to 75 years, who are citizens of the Republic of Kazakhstan;
* Patients with a clinically and laboratory confirmed diagnosis of MAFLD, without severe concomitant diseases;
* Patients who do not receive other adjuvant therapy (metabolic therapy drugs, essential phospholipids, ursodeoxycholic acid, glycyrrhizic acid, ademetionine and others);
* Patients who have at least a 7-day gap between the end of other adjuvant therapy and the start of COC and BDD;
* Patients who voluntarily signed the informed consent form.

Exclusion Criteria:

* Patients who abuse alcohol according to the AUDIT-c questionnaire;
* Patients taking COC for more than 4 weeks before signing the informed consent;
* Patients with contraindications to COC;
* Patients diagnosed with diabetes mellitus;
* Pregnancy and lactation;
* Simultaneous use of levodopa, altretamine, cisplatin, statins;
* Patients with coinfection with HIV, HBV, HCV;
* Decompensated liver cirrhosis CPT≥7 points;
* GFR ≤ 15 ml/min/1.73 m2;
* Drug-induced liver damage;
* Taking narcotic and psychotropic drugs;
* Malignant formations of the liver and other organs (in history and currently) or a clinically significant increase in alpha-fetoprotein more than >5 times;
* patients with pronounced biochemical activity (ALT, AST more than 10 ULN) and total bilirubin more than 2 ULN;
* Participation in an interventional clinical trial.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Persons aged ≥18 to 75 years inclusive with a diagnosis of metabolic-associated fatty liver disease who are undergoing outpatient monitoring at the place of residence.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-02-08 (Estimated); Study Completion 2025-02-08 (Estimated)

PRIMARY OUTCOMES:
Normalization of ALT levels during pathogenetic therapy for MAFLD at 12 months among study participants taking and not taking carnitine-orotate complex(COC) and biphenyl dimethyl dicarboxylate(BDD) | at 12 months

SECONDARY OUTCOMES:
Normalization of ALT levels during pathogenetic therapy for MAFLD at 6 months among study participants taking and not taking COC and BDD | at 6 months
Fibrosis level during pathogenetic therapy for MAFLD at 6 and 12 months among study participants taking and not taking COC and BDD | at 6 and 12 months
Steatosis level during pathogenetic therapy for MAFLD at 6 and 12 months among study participants taking and not taking COC and BDD | at 6 and 12 months
Assessment of adherence to COC and BDD therapy against the background of pathogenetic therapy for MAFLD in a cohort taking COC and BDD | up to 12 months since enrollment
Assessment of the impact of COC and BDD against the background of pathogenetic therapy for MAFLD on the quality of life of study participants taking and not taking COC and BDD | up to 12 months since enrollment
Absolute and relative risks calculation of cardiovascular diseases developing when taking COC and BDD against the background of pathogenetic therapy for MAFLD, as well as comparison among study participants taking and not taking COC and BDD | up to 12 months since enrollment
Absolute and relative risks calculation of type 2 diabetes mellitus developing when taking COC and BDD against the background of pathogenetic therapy for MAFLD, as well as comparison among study participants taking and not taking COC and BDD | up to 12 months since enrollment
Dynamics of carbohydrate metabolism parameters against the background of pathogenetic therapy for MAFLD among study participants taking and not taking COC and BDD | up to 12 months since enrollment
Dynamics of lipid metabolism parameters against the background of pathogenetic therapy for MAFLD among study participants taking and not taking COC and BDD | up to 12 months since enrollment
Frequency of registration of adverse and serious unexpected adverse events associated with the use of COC and BDD | up to 12 months since enrollment

CONTACTS AND LOCATIONS:
Locations (7):
- Kazakhstan (7):
  - State-owned public enterprise with the right of economic management "Enbekshikazakh Interdistrict Multidisciplinary Hospital", Esik, Almaty Region
  - LLP "InkarMed", Aktobe
  - hepatology center on the basis of the State Public Enterprise at the RV "City Clinic No. 5", Almaty
  - Medical Center "iClinic", Astana
  - Non-profit joint-stock company "Semey Medical University", Semey
  - Medical center "Gatromed", Shymkent
  - State-owned public enterprise with the right of economic management "Regional Clinical Hospital" of the Department of Public Health of the Turkestan region, Turkestan